CLINICAL TRIAL: NCT04408573
Title: Effects of Cycling Deep Brain Stimulation on Parkinson's Disease Gait
Brief Title: Cycling Deep Brain Stimulation on Parkinson's Disease Gait
Acronym: DBS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Rubens Gisbert Cury, Principal Investigator, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 67914017.6.0000.0068
Record Dates: First submitted 2020-05-25; First posted 2020-05-29 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: 2 weeks of regular continuous high frequency (>130Hz) stimulation, 2 weeks of cycling high frequency (>130Hz) stimulation (40sec on, 2sec off), 2 weeks of low-frequency (80Hz) continuous stimulation and 2 weeks of cycling low frequency (80Hz) stimulation (40sec on, 2sec off)
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Regular Continuous High Frequency (No Intervention): Patient remains 2 weeks in the currently chosen stimulation protocol.
- Cycling High Frequency (Experimental): Patient is stimulated with the same polarity, voltage/current, pulse width and frequency as the currently chosen stimulation protocol, but with cycling stimulation: 40sec On - 02 sec OFF
  Interventions: Other: Cycling deep brain stimulation
- Continuous Low Frequency (Experimental): Patient is stimulated with the same polarity and pulse width as the currently chosen stimulation protocol, but with low frequency (80Hz). Voltage/current will be adjusted to maintain TEED similar to that on the regular stimulation protocol.
  Interventions: Other: Cycling deep brain stimulation
- Cycling Low Frequency (Experimental): Patient is stimulated with the same polarity and pulse width as the currently chosen stimulation protocol, but with low frequency (80Hz) and cycling stimulation: 40sec On - 02 sec OFF. Voltage/current will be adjusted to maintain TEED similar to that on the regular stimulation protocol.
  Interventions: Other: Cycling deep brain stimulation

INTERVENTIONS:
Other: Cycling deep brain stimulation — Deep Brain Stimulation applied in cycling - periods of stimulation ON intercalated with periods of stimulation OFF
  Arms: Continuous Low Frequency; Cycling High Frequency; Cycling Low Frequency

SUMMARY:
Our hypothesis is that cycling DBS stimulation would be superior or non-inferior to regular DBS stimulation in Parkinson's disease patients with gait impairment. The objective of this study is compare gait disorders in patients with Parkinson's disease and DBS in 4 different scenarios: 1) regular continuous high frequency (>130Hz) stimulation, 2) cycling high frequency (>130Hz) stimulation (40sec on, 2sec off), 3) low-frequency (80Hz) continuous stimulation and 4) cycling low frequency (80Hz) stimulation (40sec on, 2sec off)

DETAILED DESCRIPTION:
Gait disorders such as falls, freezing of gait, reduction of speed, shuffling, and multi-stepped turning are common in patients with moderate and advanced Parkinson's disease. Compared to appendicular symptoms (bradykinesia, tremor, and rigidity), gait disorders tend to be more resistant to medical and regular deep brain stimulation treatment, and greatly impairs patients' quality of life and daily living activities. Some stimulation strategies have been tried to improve gait in Parkinson's disease patients, but so far most of them resulted in concomitant worsening of appendicular symptoms. However, new stimulation strategies such as cycling stimulation can potentially improve gait disorders without impairment of appendicular symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's disease
* Currently receiving Deep Brain Stimulation as a Parkinson's disease treatment
* Hoehn & Yahr stage between 2-4 during off-medication
* Underlying gait disorders despite optimal medical and stimulation treatment: score over or equal to 1 in the subitem 2.12 of the MDS-UPDRS scale
* Willingness to comply with all study procedures

Exclusion Criteria:

* Active moderate/severe psychiatric condition
* Active infection or other uncontrolled moderate/grave comorbidities
* Treatment with experimental drug
* Pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-06-19 (Actual); Primary Completion 2021-05-29 (Estimated); Study Completion 2021-12-29 (Estimated)

PRIMARY OUTCOMES:
Change in the part II of the Unified Parkinson's disease rating scale | Baseline + after 2 weeks + after 4 weeks + after 6 weeks
  The part II of the Unified Parkinson's disease rating scale (UPDRS II) is a self-reportable questionnaire consisting of 13 items that measure functionality (motor experiences of daily living). Scores vary from 0 - 52. Higher scores mean a worse outcome.
Change in the New Freezing of Gait Questionnaire | Baseline + after 2 weeks + after 4 weeks + after 6 weeks
  The New Freezing of Gait Questionnaire (NFOG-Q) is a self-reportable questionnaire consisting of 9 items that measure freezing of gait (FOG). Scores vary from 0 - 28. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Change in Falls Efficacy Scale | Baseline + after 2 weeks + after 4 weeks + after 6 weeks
  The Falls Efficacy Scale (FES) is a sixteen-item test rated on a 10-point scale from not confident at all to completely confident. It is correlated with difficulty getting up from a fall and level of anxiety. Scores vary from 16 - 64. Higher scores mean a worse outcome.
Change in The Parkinson's Disease Questionnaire (PDQ-39) | Baseline + after 2 weeks + after 4 weeks + after 6 weeks
  This questionnaire assesses how often people affected by Parkinson's experience difficulties across 8 dimensions of daily living. The 39 item questionnaire offers a patient reported measure of health status and quality of life and is the most frequently used disease-specific health status measure.Scores vary from 0 - 156. Higher scores mean a worse outcome.
Change in Activities-Specific Balance Confidence Scale (ABC scale) | Baseline + after 2 weeks + after 4 weeks + after 6 weeks
  The ABC scale is a self-report measure of balance in performing various activities without losing balance or experiencing a sense of unsteadiness. Scores vary from 0 - 100. Higher scores mean a better outcome.
Number of falls | Baseline + after 2 weeks + after 4 weeks + after 6 weeks
  Patients will be questioned about number of times they experienced falls in the last 2 weeks. Higher numbers mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Rubens G Cury, MD, PhD, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina da USP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Time Frame: Data will be made available indefinitely upon reasonable request from other authors
Access Criteria: Investigator Rubens Cury will analyse request and decide upon reasonability